CLINICAL TRIAL: NCT02684747
Title: Detecting Autologous Transfusion by Measuring Alterations in the Dynamics of Red Blood Cell Maturation and Recycling
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Sports Medicine Research and Testing Laboratory (Industry); Partnership for Clean Competition (Other)
Responsible Party: Principal Investigator, Daniel Cushman, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 83533
Record Dates: First submitted 2016-01-27; First posted 2016-02-18 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Blood Transfusion, Autologous; Blood Doping
Keywords: Healthy Volunteers; Sports Medicine; Athletes; Anti-doping
MeSH Terms: interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment - Autologous Transfusion (Experimental): Participants will be randomized to the treatment group (autologous transfusion)
  Interventions: Other: Autologous Transfusion
- Control - Normal Saline (Placebo) (Placebo Comparator): Participants will either be randomized to the control group (saline transfusion)
  Interventions: Other: Control - Normal Saline (Placebo)

INTERVENTIONS:
Other: Autologous Transfusion — Participants will receive autologous transfusion on Day 21
  Arms: Treatment - Autologous Transfusion
Other: Control - Normal Saline (Placebo) — Participants will receive saline on Day 21
  Arms: Control - Normal Saline (Placebo)

SUMMARY:
A total of 40 subjects will be recruited for participation in this study. 20 subjects (10 males and 10 females) will be randomized to the active group (those receiving re-infusion of autologous blood) and 20 subjects (10 males and 10 females) will be randomized to the placebo group (receiving NS infusion).

DETAILED DESCRIPTION:
Autologous blood transfusion is a major problem in a wide range of competitive sports. Methods with increased sensitivity, specificity, and feasibility are needed to identify athletes who cheat in this manner and compromise their health and the integrity of their sports in general. Complete blood counts (CBC) offer routine high-resolution assessment of the current hematologic status of individuals, providing estimates of a number of blood characteristics, such as the total hemoglobin concentration in the blood (HGB) and the volume fraction of cells in the blood (HCT). These CBC components are homeostatically controlled by the carefully regulated dynamic processes of red blood cell (RBC) production in and release from the bone marrow, RBC maturation in the peripheral circulation over the course of the ~100-day RBC lifespan, and clearance and recycling of senescent cells. Any significant perturbation to the circulating population of RBCs, like autologous transfusion, will immediately trigger compensatory modulation of one or more of these dynamic processes. The investigators believe quantification of these underlying dynamic processes will enable us to detect autologous transfusion. These dynamic RBC processes cannot currently be measured directly, but novel mathematical modeling enables their inference from routine complete blood and reticulocyte counts. The investigators propose to test the ability of modeled RBC dynamics to identify instances of autologous blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18-35 years old
2. Classified as low risk and will not have any major signs or symptoms suggestive of cardiovascular, pulmonary, or metabolic disease according to the American College of Sports Medicine's (ACSM) risk stratification categories
3. The subjects should be well-trained endurance athletes. This group could consist of cyclists (road and mountain), triathletes, runners, long-distance swimmers, etc.

Exclusion Criteria:

1. Age less than 18 or greater than 35 on the day of enrollment
2. Any contraindication to blood donation as defined by the American Association of Blood Banks http://www.fda.gov/downloads/BiologicsBloodVaccines/BloodBloodProducts/QuestionsaboutBlood/UCM272981.pdf
3. Any chronic illness (e.g.diabetes, heart disease, hypotension, anemia, hemoglobinopathy, marrow diseases, leukemia/lymphoma, pregnancy, amenorrhea/female athlete triad)
4. Any abnormal CBC index or iron study; any blood dyscrasia
5. Abnormal blood and urine tests for doping agents (e.g. phthalates)
6. Positive uhCG or women who are attempting to get pregnant during the study period
7. Unwilling or unable to provide blood samples or receive a blood transfusion
8. Not a participant in endurance sports activities
9. Are currently on any medications that might affect hematologic parameters including, but not restricted to, hematopoietic medications
10. Subjects with a baseline hemoglobin above 16.7 g/dL, or baseline hematocrit below 35% or above 55%.
11. Any subject that plans to participate in an organized athletic event (or USA Cycling sanctioned event) within 30 days following the re-infusion phase of the study will not be allowed to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Hematocrit | 8 weeks
  This will be used within a mathematical model to define the volume (v) and hemoglobin (h) dynamics of a typical RBC as deterministic functions (f) and random fluctuations in the rates of these changes over time (ζ) (Patel, Patel, & Higgins, 2015).
Hemoglobin | 8 weeks
  This will be used within a mathematical model to define the volume (v) and hemoglobin (h) dynamics of a typical RBC as deterministic functions (f) and random fluctuations in the rates of these changes over time (ζ) (Patel, Patel, & Higgins, 2015).
Reticulocyte count | 8 weeks
  This will be used within a mathematical model to define the volume (v) and hemoglobin (h) dynamics of a typical RBC as deterministic functions (f) and random fluctuations in the rates of these changes over time (ζ) (Patel, Patel, & Higgins, 2015).
Mean corpuscular volume | 8 weeks
  This will be used within a mathematical model to define the volume (v) and hemoglobin (h) dynamics of a typical RBC as deterministic functions (f) and random fluctuations in the rates of these changes over time (ζ) (Patel, Patel, & Higgins, 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cushman, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Center for Clinical & Translational Science, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cowell HR, Swickard JW. Autotransfusion in children's orthopaedics. J Bone Joint Surg Am. 1974 Jul;56(5):908-12. No abstract available. PMID 4847238
- [Background] Cregan P, Donegan E, Gotelli G. Hemolytic transfusion reaction following transfusion of frozen and washed autologous red cells. Transfusion. 1991 Feb;31(2):172-5. doi: 10.1046/j.1537-2995.1991.31291142950.x. PMID 1996486
- [Background] Domen RE. Adverse reactions associated with autologous blood transfusion: evaluation and incidence at a large academic hospital. Transfusion. 1998 Mar;38(3):296-300. doi: 10.1046/j.1537-2995.1998.38398222875.x. PMID 9563411
- [Background] Higgins JM, Mahadevan L. Physiological and pathological population dynamics of circulating human red blood cells. Proc Natl Acad Sci U S A. 2010 Nov 23;107(47):20587-92. doi: 10.1073/pnas.1012747107. Epub 2010 Nov 8. PMID 21059904
- [Background] Kumar S, Goyal K, Dube SK, Dubey S, Bindra A, Kedia S. Anaphylactic reaction after autologous blood transfusion: A case report and review of the literature. Asian J Neurosurg. 2015 Apr-Jun;10(2):145-7. doi: 10.4103/1793-5482.154983. PMID 25972952
- [Background] Morkeberg J, Belhage B, Ashenden M, Borno A, Sharpe K, Dziegiel MH, Damsgaard R. Screening for autologous blood transfusions. Int J Sports Med. 2009 Apr;30(4):285-92. doi: 10.1055/s-0028-1105938. Epub 2009 Feb 6. PMID 19199200
- [Background] Popovsky MA, Whitaker B, Arnold NL. Severe outcomes of allogeneic and autologous blood donation: frequency and characterization. Transfusion. 1995 Sep;35(9):734-7. doi: 10.1046/j.1537-2995.1995.35996029156.x. PMID 7570932
- [Background] Pottgiesser T, Sottas PE, Echteler T, Robinson N, Umhau M, Schumacher YO. Detection of autologous blood doping with adaptively evaluated biomarkers of doping: a longitudinal blinded study. Transfusion. 2011 Aug;51(8):1707-15. doi: 10.1111/j.1537-2995.2011.03076.x. Epub 2011 Mar 7. PMID 21382045
- [Background] Solymos E, Guddat S, Geyer H, Flenker U, Thomas A, Segura J, Ventura R, Platen P, Schulte-Mattler M, Thevis M, Schanzer W. Rapid determination of urinary di(2-ethylhexyl) phthalate metabolites based on liquid chromatography/tandem mass spectrometry as a marker for blood transfusion in sports drug testing. Anal Bioanal Chem. 2011 Aug;401(2):517-28. doi: 10.1007/s00216-010-4589-4. Epub 2010 Dec 25. PMID 21188579
- [Background] Weatherall DJ. Systems biology and red cells. N Engl J Med. 2011 Jan 27;364(4):376-7. doi: 10.1056/NEJMcibr1012683. No abstract available. PMID 21268732
- [Background] Basson, M. Red blood cells by the numbers. Nature Medicine 16, 1 (2010).